CLINICAL TRIAL: NCT02019251
Title: Evaluation of Regional Lung Function in Lung Transplant Recipients Using 19F Magnetic Resonance Imaging of Inert Perfluorinated Gases Mixed With Oxygen
Brief Title: Lung Transplant Subjects Using 19F MRI
Acronym: DIAL1001005
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hal C Charles (Other)
Responsible Party: Sponsor-Investigator, Hal C Charles, Associate Professor Department of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00047929; DIAL1001005 (Other: Duke University Medical Center)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Post Single or Double Lung Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Post single or double lung transplant (Experimental): The subjects will receive the gas by breathing perfluorinated gas/oxygen mixture using Disposable Face mask and a standard Douglas Bag system.
  Interventions: Drug: perfluorinated gas/oxygen mixture; Device: MRI

INTERVENTIONS:
Drug: perfluorinated gas/oxygen mixture — Subjects are imaged with MRI one time with the use of perfluorinated gas / oxygen mixtures as an MRI contrast agent for lung function.
Device: MRI

SUMMARY:
The goal of this study is to evaluate the utilization of conventional 'thermally' polarized perfluorinated gases mixed with oxygen as inhaled inert contrast agents to image the airway spaces in subjects who have undergone single or double lung transplantation. This is an open label study expanding on current work here at Duke. Images will be obtained using 19F MRI during wash-in and washout for evaluation of ventilation efficiency.

DETAILED DESCRIPTION:
This is an open label study in up to 10 lung transplant recipients post lung transplantation whose post-transplant status is being monitored according to local standard of care. Each subject will receive up to 20 liters of PFP/oxygen gas mixtures as a contrast agent to visualize the airway and alveolar spaces in their lungs using 19F magnetic resonance imaging of inert gas/oxygen mixtures.

The goal of this study is to evaluate the utilization of conventional 'thermally' polarized perfluorinated gases mixed with oxygen as an exogenous inert contrast agent to image the airway spaces in subjects with transplanted lungs. This is an open label proof of concept study expanding on work here at Duke.

The central hypothesis and current observation is that PFx gases, when used as contrast agents, provide functional images of the lung airways including important regional ventilation information such as ventilation defect severity and gas trapping. We will test the central hypothesis and accomplish the overall objective by addressing the following specific aims:

Primary Study Aims/Secondary Aims Aim 1: Determine qualitative and quantitative measures of lung ventilation performance in terms of ventilation efficiency during wash-in evaluation of the 19F images of lung airspaces.

Aim 2: Determine qualitative and quantitative measures of lung ventilation performance in terms of direct measures of gas trapping measured during washout of the perfluorinated gas mixture.

The outcomes of the work proposed in the aims is expected to demonstrate a non-invasive novel quantitative approach for evaluation of regional lung function in subjects with lung transplants that would allow repeated evaluation of lung function post-transplant to monitor for chronic allograft rejection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:
* Subjects must be ≥ 18 years of age;
* Post single or double lung transplant;
* Subjects who are willing and able to comply with scheduled visits and other trial procedures

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the trial:
* Unable to undergo a 3.0-Tesla MRI exam of the lungs and chest because of contraindications (e.g. metal in the eye, claustrophobia);
* Unable to receive gas mixture by breathing because of contraindications;
* Participation in a clinical trial with a study drug that may impact lung function in the past 14 days; or
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
* Female; women at risk of pregnancy are required to have a confirmed negative blood pregnancy test at Screening if of childbearing potential prior to the MRI scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
obtain regional, non-invasive images of pulmonary function in patient's post lung transplantation | 1 day (Single exposure)

CONTACTS AND LOCATIONS:
Overall Officials: Cecil Charles, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States